CLINICAL TRIAL: NCT05693701
Title: Implementing a Multicomponent Intervention to Treat Blood Donors With Familial Hypercholesterolemia
Brief Title: Multicomponent Intervention Study- Blood Donors With High Cholesterol
Acronym: DONATE-FH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Amit Khera, PROFESSOR - Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STU-2020-1366; 1R61HL161753-01 (NIH)
Record Dates: First submitted 2023-01-11; First posted 2023-01-23 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Lipid Metabolism Disorder
Keywords: Blood Donors; High Cholesterol; LDL Cholesterol
MeSH Terms: conditions — Lipid Metabolism Disorders; Hypercholesterolemia

STUDY DESIGN:
Intervention Model Description: Treatment assignment will be via block randomization stratified on age category in a 1:1 allocation ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Usual care) (Other): This arm will receive standard notification that is usually provided by Carter describing need to review with donor's primary care physician the presence of high cholesterol
  Interventions: Other: Usual care notification
- Intervention Group (Implementation strategy bundle) (Experimental): Along with standard high cholesterol notification from Carter BloodCare, this arm will receive Implementation strategy bundle (educational material regarding high cholesterol levels)
  Interventions: Behavioral: Implementation Strategy Bundle; Other: Usual care notification

INTERVENTIONS:
Behavioral: Implementation Strategy Bundle — Bundle includes multimodal communications to notify donors about high cholesterol and its treatment, website with resources, and an optional care navigator. Resources for their primary care provider will also be disseminated.
  Arms: Intervention Group (Implementation strategy bundle)
Other: Usual care notification — Carter BloodCare will notify participants of their high cholesterol, potential for genetic causes, and recommendation to see their care provider by sending its routine, standard notification letter. These participants will also be eligible to receive the intervention bundle at the end of the study.

SUMMARY:
The purpose and objective of this study is to improve cholesterol treatment among blood donors with FH (Familial Hypercholesterolemia).

DETAILED DESCRIPTION:
This is a single center randomized, two arm trial. The two study arms include usual care (standard notification) and implementation bundle intervention. UT Southwestern Medical Center will be the main study site and Carter Blood Care will serve as the recruitment site.

Screening/Baseline visit: Donors agreeing to participate in the study will be informed of study procedures and will provide informed consent. A 20 mL blood sample as well as a urine sample will be obtained for eligibility screening laboratories and baseline LDL-C.

Follow-up phone call: At 3 months post-randomization, participants in both arms will be briefly contacted by phone by the Research Assistant to thank them for their participation and to answer any study related questions.

End of study 6 month visit. Participants will engage in a virtual visit for end of study procedures. At this follow-up visit, the Research Assistant will assess for any adverse events and direct the participant to collect a fasting blood sample for repeat LDL-C measurement. The Research Assistant will administer an electronic survey and knowledge questionnaires. Additional clinical visits as desired by the participants' physicians will be allowed at their discretion.

ELIGIBILITY:
Inclusion Criteria:

* Blood donors from Carter BloodCare with high cholesterol meeting MEDPED FH criteria
* Age 18 to 75 years

Exclusion Criteria:

* Currently taking medication to lower cholesterol
* Taking any medication that can interact with statins
* Pregnancy
* Identified secondary cause of elevated lipids
* Chronic liver disease or significantly elevated liver function tests (> 3 times upper limit)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Difference in change in LDL cholesterol levels from baseline to 6 months | Baseline, 6 months
  This is the difference between the two study arms in change in LDL cholesterol level measurements obtained from lab work of blood samples from baseline and at 6 months

SECONDARY OUTCOMES:
Difference in 6 month LDL-C values between the two treatment arms | 6 months
  This is the difference between the two study arms in the 6 month LDL cholesterol levels obtained from lab work of blood samples.
Proportion of participants prescribed high-intensity statin therapy | 6 months
  Proportion of participants prescribed high-intensity statin therapy will be calculated as the number of patients who were prescribed high-intensity statin therapy in each arm divided by the total number of participants analyzed in each arm
Proportion of participants prescribed any statin therapy | 6 months
  Proportion of participants prescribed any statin therapy will be calculated as the number of patients who were prescribed any statin therapy in each arm divided by the total number of participants analyzed in each arm
Difference in participants' knowledge regarding FH at the end of study | 6 months
  Difference in participant's knowledge regarding FH at 6 months is measured using a validated FH knowledge survey where higher scores indicate greater knowledge. Comparisons between the two study arms will be made.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Khera, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No